CLINICAL TRIAL: NCT02382887
Title: Comparison by Neuromonitoring of Two Techniques of Tracheal Intubation in Patients With Unstable Cervical Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Patrick Schoettker,MD PD, MD, PD, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 225/08
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Spinal Injuries
Keywords: intubation; difficult airway; fiberscopy; Airtraq; general anesthesia
MeSH Terms: conditions — Spinal Injuries | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tracheal intubation with Fiberscopy (Active Comparator): tracheal intubation with a fiberscope
  Interventions: Procedure: tracheal intubation; Device: fiberscope
- Tracheal intubation with Airtraq (Experimental): tracheal intubation with an Airtraq
  Interventions: Procedure: tracheal intubation; Device: Airtraq

INTERVENTIONS:
Procedure: tracheal intubation — tracheal intubation with the Airtraq
Device: Airtraq
  Arms: Tracheal intubation with Airtraq
Device: fiberscope
  Arms: Tracheal intubation with Fiberscopy

SUMMARY:
Patients who present with an unstable cervical spine following an accident need a general anesthesia for the necessary surgery.

Commonly, the management of the tracheal intubation is performed by a fiberoptic technique.

However, changes in equipment availability and quality may challenge the fiberoptic intubation technique.

The investigators wish to compare the tracheal intubations performed with the Airtraq in comparison with the fiberscopic technique.

DETAILED DESCRIPTION:
Patients who present with an unstable cervical spine following an accident need a general anesthesia for the necessary surgery.

Commonly, the management of the tracheal intubation is performed by a fiberoptic technique (historic gold standard technique).

However, changes in equipment availability and quality may challenge the fiberoptic intubation technique.

We wish to compare the tracheal intubations performed with the Airtraq in comparison with the fiberscopic technique.

Primary outcomes will be the changes in neurophysiologic responses monitored by a neurophysiologist in 5 specific phases:

1. Basal potential (BM): neuromonitoring while the patient is anesthetized, no movements
2. Ventilation potential (VM): neuromonitoring while the patient is anesthetized and a bag-mask ventilation is performed
3. Intubation potential (IP): neuromonitoring while the patient is being intubated with one of the two randomized devices
4. Post Intubation (PI): neuromonitoring after the patient has been intubated
5. Post Positioning (PP): neuromonitoring after the patient has been properly positioned on the operating table and is ready for surgery

ELIGIBILITY:
Inclusion Criteria:

* unstable cervical spine due to a cervical vertebra fracture
* American Society of Anesthesia classification 1-3
* BMI < 30 kg/m2
* patients necessitating a general anesthesia for surgery

Exclusion Criteria:

* patient refusal
* ASA >3
* mouth opening < 15mm
* patients with known history of previous orotracheal tumor surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Neuromonitoring modifications (modifications appearing on the neuromonitoring) | 30 seconds
  modifications appearing on the neuromonitoring during the 5 different phases

SECONDARY OUTCOMES:
time necessary for tracheal intubation | 180 seconds
tracheal inlet view (best view during intubation) | 10 seconds
  best view during intubation
number of attempts necessary | 180 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoettker, MD, PD, Principal Investigator — Chief Medical Officer
Locations (1):
- Dpt of Anesthesiology, University of Lausanne CHUV, Lausanne, Canton of Vaud, Switzerland